CLINICAL TRIAL: NCT07260149
Title: Coordinated Care for Alcohol Problems (CCAP): a Randomised Controlled Trial From Goa, India
Brief Title: Coordinated Care for Alcohol Problems
Acronym: CCAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sangath (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AN_2025_119
Record Dates: First submitted 2025-11-16; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol use disorder; Coordinated care; Complex intervention; Digital intervention; Psychosocial intervention; Non-specialist health workers; Task-sharing; Randomised controlled trial; India
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CCAP (Experimental): Hazardous drinking: M-BIT is an eight-week digital intervention delivered over WhatsApp.
  Harmful drinking: CAP is a manualised brief psychological treatment for harmful drinking. CAP+ will include treatment engagement strategies integrated into CAP.
  Dependent drinking: CONTAD is a manualised treatment comprising of 5-7 days of supervised home detoxification followed by relapse prevention counselling for dependent drinking.
  Participants with harmful and dependent drinking level will be offered referral to the public District Hospitals or the state Psychiatric Hospital for assessment of eligibility for anti-craving medicines if available and to be prescribed and dispensed as per their Standard Operating Procedures.
  Interventions: Behavioral: CCAP
- Enhanced usual care (Active Comparator): Hazardous drinking: Brief intervention leaflet which is an information sheet/brochure with information on alcohol consumption, associated risks, and tips to manage and reduce drinking.
  Harmful drinking: CAP is a manualised brief psychological treatment for harmful drinking. It has three phases which are delivered in one to four sessions over six to eight weeks by NSHWs. Each session lasts between 30 to 45 minutes. The content is delivered through motivational interviewing with additional behavioural and cognitive components. CAP has proven to be effective and cost-effective in reducing drinking in men with harmful level of drinking in a prior study. CAP can be delivered in any of the local vernacular (Hindi, Marathi, Konkani) or English.
  Dependent drinking: Supported in-patient detoxification which is hospital-based detoxification delivered in secondary or tertiary care.
  Interventions: Behavioral: Enhanced usual care

INTERVENTIONS:
Behavioral: CCAP — Hazardous drinking: The content of the intervention includes seven themes: health education, alcohol reduction, drinking and risk management, drinking alternatives, situational content, urge management, and relapse prevention. Participants will receive texts and video-based messages building their awareness about drinking and associated harms.
  Harmful drinking: CAP has three phases which are delivered in one to four sessions over six to eight weeks by NSHWs. Each session lasts between 30 to 45 minutes. The content is delivered through motivational interviewing with additional behavioural and cognitive components. CAP+ will include treatment engagement strategies integrated into CAP.
  Dependent drinking: Home detoxification will be supervised by a doctor and monitored by the NSHW and a designated carer (e.g. spouse) for the patient at their home-setting. The counselling sessions are delivered by NSHWs, over 4-8 weeks and lasting 30-60 minutes each.
  Arms: CCAP
Behavioral: Enhanced usual care — Hazardous drinking: An information sheet/brochure with information on alcohol consumption, associated risks, and tips to manage and reduce drinking.
  Harmful drinking: CAP psychological brief treatment delivered by trained NSHWs (described above in detail).
  Dependent drinking: Hospital-based detoxification delivered in secondary or tertiary care.
  Arms: Enhanced usual care

SUMMARY:
Parallel group individually randomised controlled trial (RCT) with stratified (by severity of drinking problem) randomisation into intervention and control arms. Aim is to test the effectiveness and cost-effectiveness of Coordinated Care for Alcohol Problems (CCAP) for the whole spectrum of drinking problems in primary care in Goa, India. Primary outcome is the drinking outcome of percentage days abstinent (PDA) at three months post randomisation. Secondary outcomes include drinking outcomes (PDA at six- and 12- months post-randomisation; percentage days heavy drinking (PDHD), intensity of drinking and remission) and drinking related outcomes (e.g., injuries, violence) at three-, six- and 12- months post- randomisation. Participants will include consenting adult (>18 years) men with drinking problems attending Primary Healthcare Centres (PHCs) and Community Healthcare Centres (CHCs) in Goa and have drinking problems defined as scoring >8 on the Alcohol Use Disorder Identification Test (AUDIT). CCAP is a multi-component evidence-informed complex intervention package for coordinating treatment for all levels of problem drinking (hazardous, harmful, dependent). For hazardous drinking, it includes Mobile based Brief Intervention Treatment (M-BIT), which is a mobile-messaging brief intervention delivered via WhatsApp over eight weeks using multimedia content including contextually relevant messages, images and videos. For harmful drinking, it includes Counselling for Alcohol Problems Plus (CAP+) which is Counselling for Alcohol Problems (CAP), an evidence-based brief psychological treatment, integrated with strategies to enhance treatment engagement (entry into and completion). For dependent drinking, it includes Community Orientated Treatment for Alcohol Dependence (CONTAD) which is supervised home-detoxification over a week followed by a psychological treatment to prevent relapse, both integrated with treatment engagement strategies. CAP+ and CONTAD will be delivered in the community by non-specialist health workers (NSHW).

ELIGIBILITY:
Inclusion Criteria:

1. Scoring positive for problem drinking (≥ 8 on the AUDIT)
2. Have been residing in Goa for more than 12 continuous preceding months as an indicator of stability of residence which would be required both for treatment delivery and completion of outcome evaluation.
3. Language:

   1. For hazardous drinking (AUDIT score of 8-15), patients must be able to understand at least one of the local vernacular languages (Hindi or Konkani) or English. Patients must be able to read at least one of the local vernacular languages (Hindi or Marathi) or English.
   2. For harmful and dependent drinking (AUDIT score of >15), patients must be able to understand and speak any of the local vernacular languages (Konkani, Marathi, Hindi) or English.
4. For hazardous drinking, patients must also have access to a personal smartphone with WhatsApp.
5. For dependent drinking (AUDIT score of >19), patients must consent for home visits and must also be eligible for home detoxification as per structured detoxification protocol.

Exclusion Criteria:

1. For hazardous drinking, patients with significant visual or hearing impairment will be ineligible due to the audio-visual nature of the intervention.
2. For harmful and dependent drinking, patients with significant speech, hearing, or language impairment (as evident during screening) will be excluded as the intervention is primarily a 'talking treatment'.
3. For patients who present to the PHC/CHC needing urgent medical attention (emergency treatment or in-patient admission), screening will be deferred until their condition is stable.
4. Those who are alcohol dependent and do not meet the eligibility criteria for home detoxification as per protocol.
5. Those who are alcohol dependent but are currently not drinking. As AUDIT covers a period of 12 months, it will also detect those who meet the criteria for alcohol dependence over the past 12 months but are currently abstinent (hence not eligible for detoxification).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1022 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage days abstinent (PDA) [Parent trial] | 3 months post randomisation
  Proportion of days abstinent in the past two weeks measured using the Timeline Follow Back (TLFB)
Pattern of drinking [Sub-group A Hazardous drinking] | 3 months post randomisation
  Number of heavy drinking days in the past two weeks measured using the TLFB
Treatment completion [Sub-group B Harmful Drinking] | Through the period of intervention delivery, an average of 3 months
  Proportion of consented participants who go on to complete treatment defined as planned discharge which would be one of the following
  1. Received all sessions as per protocol
  2. Discharge by mutual agreement between NSHW and participant on achievement of treatment goals
  3. Referral out of the study
Intensity of drinking [Sub-group C Dependent drinking] | 3 months post randomisation
  Units of alcohol consumed in the past week measured using the TLFB

SECONDARY OUTCOMES:
Percentage days abstinent (PDA) [Parent trial] | 6 months post randomisation
  Proportion of days abstinent in the past two weeks measured using the Timeline Follow
Percentage days abstinent (PDA) [Parent trial] | 12 months post randomisation
  Proportion of days abstinent in the past two weeks measured using the Timeline Follow
Consequences of alcohol use [Parent trial] | 3 months post randomisation
  Physical, social, intrapersonal and interpersonal consequences of alcohol use measured using the Short Inventory of Problems (SIP)
Consequences of alcohol use [Parent trial] | 6 months post randomisation
  Physical, social, intrapersonal and interpersonal consequences of alcohol use measured using the Short Inventory of Problems (SIP)
Consequences of alcohol use [Parent trial] | 12 months post randomisation
  Physical, social, intrapersonal and interpersonal consequences of alcohol use measured using the Short Inventory of Problems (SIP)
Food security [Parent trial] | 12 months post randomisation
  Improvement of food security as measured using Food Insecurity Experience Scale
Pattern of drinking [Parent trial] | 3 months post randomisation
  Percentage days heavy drinking (PDHD) in the past two weeks measured using the TLFB
Pattern of drinking [Parent trial] | 6 months post randomisation
  Percentage days heavy drinking (PDHD) in the past two weeks measured using the TLFB
Pattern of drinking [Parent trial] | 12 months post randomisation
  Percentage days heavy drinking (PDHD) in the past two weeks measured using the TLFB
Intensity of drinking [Parent trial] | 3 months post randomisation
  Grams ethanol consumed per drinking day in the past two weeks measured using the TLFB
Intensity of drinking [Parent trial] | 6 months post randomisation
  Grams ethanol consumed per drinking day in the past two weeks measured using the TLFB
Intensity of drinking [Parent trial] | 12 months post randomisation
  Grams ethanol consumed per drinking day in the past two weeks measured using the TLFB
Remission [Parent trial] | 3 months post randomisation
  Alcohol Use Disorder Identification Test (AUDIT) score <8
Remission [Parent trial] | 6 months post randomisation
  Alcohol Use Disorder Identification Test (AUDIT) score <8
Remission [Parent trial] | 12 months post randomisation
  Alcohol Use Disorder Identification Test (AUDIT) score <8
System-level costs [Parent trial] | Monthly, during the period of implementation
  Economic costs in WHO six building blocks for delivering the interventions measured using inventory form for collecting system-level economic costs of delivering interventions (finance records and individuals involved in delivery of interventions)
Out-of-pocket costs 1 [Parent trial] | 3 months post randomisation
  Out-of-pocket costs for receiving general medical care and the related non-medical costs (e.g.: time loss, travel, etc) measured using Client Service Receipt Inventory form for collecting costs to patients who receive CCAP interventions
Out-of-pocket costs 1 [Parent trial] | 6 months post randomisation
  Out-of-pocket costs for receiving general medical care and the related non-medical costs (e.g.: time loss, travel, etc) measured using Client Service Receipt Inventory form for collecting costs to patients who receive CCAP interventions
Out-of-pocket costs 1 [Parent trial] | 12 months post randomisation
  Out-of-pocket costs for receiving general medical care and the related non-medical costs (e.g.: time loss, travel, etc) measured using Client Service Receipt Inventory form for collecting costs to patients who receive CCAP interventions
Out-of-pocket costs 2 [Parent trial] | 3 months post randomisation
  Out-of-pocket costs for receiving CCAP interventions (e.g.: time loss, travel, etc) using survey form for receiving the CCAP interventions to patients who receive CCAP interventions
Out-of-pocket costs 2 [Parent trial] | 6 months post randomisation
  Out-of-pocket costs for receiving CCAP interventions (e.g.: time loss, travel, etc) using survey form for receiving the CCAP interventions to patients who receive CCAP interventions
Out-of-pocket costs 2 [Parent trial] | 12 months post randomisation
  Out-of-pocket costs for receiving CCAP interventions (e.g.: time loss, travel, etc) using survey form for receiving the CCAP interventions to patients who receive CCAP interventions
Disability [Parent trial] | 3 months post randomisation
  Standardised disability scores used to estimate Quality-Adjusted Life Years (QALYs) using the WHO Disability Assessment Scale (WHODAS)
Disability [Parent trial] | 6 months post randomisation
  Standardised disability scores used to estimate Quality-Adjusted Life Years (QALYs) using the WHO Disability Assessment Scale (WHODAS)
Disability [Parent trial] | 12 months post randomisation
  Standardised disability scores used to estimate Quality-Adjusted Life Years (QALYs) using the WHO Disability Assessment Scale (WHODAS)
Pattern of drinking [Sub-group A Hazardous drinking] | 6 months post randomisation
  Number of heavy drinking days in the past two weeks measured using the TLFB
Pattern of drinking [Sub-group A Hazardous drinking] | 12 months post randomisation
  Number of heavy drinking days in the past two weeks measured using the TLFB
Intensity of drinking [Sub-group A Hazardous drinking] | 3 months post randomisation
  Grams ethanol consumed per drinking day in past two weeks measured using the TLFB
Intensity of drinking [Sub-group A Hazardous drinking] | 6 months post randomisation
  Grams ethanol consumed per drinking day in past two weeks measured using the TLFB
Intensity of drinking [Sub-group A Hazardous drinking] | 12 months post randomisation
  Grams ethanol consumed per drinking day in past two weeks measured using the TLFB
Remission [Sub-group A Hazardous drinking] | 3 months post randomisation
  Alcohol Use Disorder Identification Test (AUDIT) score <8
Remission [Sub-group A Hazardous drinking] | 6 months post randomisation
  Alcohol Use Disorder Identification Test (AUDIT) score <8
Remission [Sub-group A Hazardous drinking] | 12 months post randomisation
  Alcohol Use Disorder Identification Test (AUDIT) score <8
Percentage days abstinent (PDA) [Sub-group A Hazardous drinking] | 3 months post randomisation
  Proportion of days abstinent in the past two weeks measured using the TLFB
Percentage days abstinent (PDA) [Sub-group A Hazardous drinking] | 6 months post randomisation
  Proportion of days abstinent in the past two weeks measured using the TLFB
Percentage days abstinent (PDA) [Sub-group A Hazardous drinking] | 12 months post randomisation
  Proportion of days abstinent in the past two weeks measured using the TLFB
Pattern of drinking [Sub-group A Hazardous drinking] | 3 months post randomisation
  Percentage days heavy drinking (PDHD) in the past two weeks measured using the TLFB
Pattern of drinking [Sub-group A Hazardous drinking] | 6 months post randomisation
  Percentage days heavy drinking (PDHD) in the past two weeks measured using the TLFB
Pattern of drinking [Sub-group A Hazardous drinking] | 12 months post randomisation
  Percentage days heavy drinking (PDHD) in the past two weeks measured using the TLFB
Treatment entry [Sub-group B Harmful drinking] | 3 months post randomisation
  Proportion of consented participants who receive at least one session of counselling
Treatment entry [Sub-group B Harmful drinking] | 6 months post randomisation
  Proportion of consented participants who receive at least one session of counselling
Treatment entry [Sub-group B Harmful drinking] | 12 months post randomisation
  Proportion of consented participants who receive at least one session of counselling
Percentage days abstinent (PDA) [Sub-group B Harmful drinking] | 3 months post randomisation
  Proportion of days abstinent in the past two weeks measured using the TLFB
Percentage days abstinent (PDA) [Sub-group B Harmful drinking] | 6 months post randomisation
  Proportion of days abstinent in the past two weeks measured using the TLFB
Percentage days abstinent (PDA) [Sub-group B Harmful drinking] | 12 months post randomisation
  Proportion of days abstinent in the past two weeks measured using the TLFB
Pattern of drinking [Sub-group B Harmful drinking] | 3 months post randomisation
  Percentage days heavy drinking (PDHD) in the past two weeks measured using the TLFB
Pattern of drinking [Sub-group B Harmful drinking] | 6 months post randomisation
  Percentage days heavy drinking (PDHD) in the past two weeks measured using the TLFB
Pattern of drinking [Sub-group B Harmful drinking] | 12 months post randomisation
  Percentage days heavy drinking (PDHD) in the past two weeks measured using the TLFB
Intensity of drinking [Sub-group B Harmful drinking] | 3 months post randomisation
  Grams ethanol consumed per drinking day in past two weeks measured using the TLFB
Intensity of drinking [Sub-group B Harmful drinking] | 6 months post randomisation
  Grams ethanol consumed per drinking day in past two weeks measured using the TLFB
Intensity of drinking [Sub-group B Harmful drinking] | 12 months post randomisation
  Grams ethanol consumed per drinking day in past two weeks measured using the TLFB
Remission [Sub-group B Harmful drinking] | 3 months post randomisation
  Alcohol Use Disorder Identification Test (AUDIT) score <8
Remission [Sub-group B Harmful drinking] | 6 months post randomisation
  Alcohol Use Disorder Identification Test (AUDIT) score <8
Remission [Sub-group B Harmful drinking] | 12 months post randomisation
  Alcohol Use Disorder Identification Test (AUDIT) score <8
Consequences of alcohol use [Sub-group B Harmful drinking] | 3 months post randomisation
  Physical, social, intrapersonal and interpersonal consequences of alcohol use measured using the Short Inventory of Problems (SIP)
Consequences of alcohol use [Sub-group B Harmful drinking] | 6 months post randomisation
  Physical, social, intrapersonal and interpersonal consequences of alcohol use measured using the Short Inventory of Problems (SIP)
Consequences of alcohol use [Sub-group B Harmful drinking] | 12 months post randomisation
  Physical, social, intrapersonal and interpersonal consequences of alcohol use measured using the Short Inventory of Problems (SIP)
Food security [Sub-group B Harmful drinking] | 12 months post randomisation
  Improvement of food security as measured using Food Insecurity Experience Scale
Intensity of drinking [Sub-group C Dependent drinking] | 6 months post randomisation
  Units of alcohol consumed in the past week measured using TLFB
Intensity of drinking [Sub-group C Dependent drinking] | 12 months post randomisation
  Units of alcohol consumed in the past week measured using TLFB
Consequences of alcohol use [Sub-group C Dependent drinking] | 3 months post randomisation
  Physical, social, intrapersonal and interpersonal consequences of alcohol use measured using the Short Inventory of Problems (SIP)
Consequences of alcohol use [Sub-group C Dependent drinking] | 6 months post randomisation
  Physical, social, intrapersonal and interpersonal consequences of alcohol use measured using the Short Inventory of Problems (SIP)
Consequences of alcohol use [Sub-group C Dependent drinking] | 12 months post randomisation
  Physical, social, intrapersonal and interpersonal consequences of alcohol use measured using the Short Inventory of Problems (SIP)
Food security [Sub-group C Dependent drinking] | 12 months post randomisation
  Improvement of food security as measured using Food Insecurity Experience Scale
Remission [Sub-group C Dependent drinking] | 3 months post randomisation
  Alcohol Use Disorder Identification Test (AUDIT) score <8
Remission [Sub-group C Dependent drinking] | 6 months post randomisation
  Alcohol Use Disorder Identification Test (AUDIT) score <8
Remission [Sub-group C Dependent drinking] | 12 months post randomisation
  Alcohol Use Disorder Identification Test (AUDIT) score <8
Treatment entry [Sub-group C Dependent drinking] | Through the period of intervention delivery, an average of 3 months
  Proportion of consented participants who receive at least one session of counselling
Treatment completion [Sub-group C Dependent drinking] | Through the period of intervention delivery, an average of 3 months
  Proportion of consented participants who go on to complete treatment defined as planned discharge which would be one of the following
  1. Received all sessions as per protocol
  2. Discharge by mutual agreement between NSHW and participant on achievement of treatment goals
  3. Referral out of the program